CLINICAL TRIAL: NCT06695832
Title: Adjunctive Fosfomycin for Treatment of Staphylococcus Aureus Bacteraemia: Protocol for a Pooled Post-hoc Analysis of Two Randomised Clinical Trials
Brief Title: Adjunctive Fosfomycin for Treatment of Staphylococcus Aureus Bacteraemia
Acronym: BACSAFO
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Francesc Escrihuela-Vidal, Medical Doctor, Hospital Universitari de Bellvitge
Other Study IDs: EOM033/24
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Staphylococcus aureus bacteremia; Fosfomycin; Daptomycin; Cloxacillin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adjunctive fosfomycin: All patients receiving adjunctive fosfomycin (the combination therapy group).
- Standard antibiotic monotherapy group: All patients not receiving fosfomycin, i.e., those receiving daptomycin alone for MRSA bacteraemia or cloxacillin alone for MSSA bacteraemia.

SUMMARY:
Staphylococcus aureus bacteraemia is a frequent and life-threatening infection, despite current standard antibiotic monotherapy. This study aims to clarify the role of fosfomycin as an adjunctive therapy for improving outcomes in patients with this serious infection. Two clinical trials suggested that adjunctive fosfomycin therapy might offer a clinical benefit in certain cases, but the results are inconclusive. We aim to analyse pooled data from these trials in order to identify subgroups of patients that might benefit most from this therapy.

DETAILED DESCRIPTION:
Background. Improving outcomes in patients with methicillin-susceptible (MSSA) and methicillin-resistant (MRSA) Staphylococcus aureus bacteraemia (SAB) is a critical healthcare goal. Two recent randomised clinical trials (RCTs), the BACSARM trial and the SAFO trial, assessed the efficacy of fosfomycin as an adjunctive therapy for MRSA and MSSA SAB respectively. Although neither trial demonstrated statistically significant differences in their primary endpoints of treatment success and reduced mortality respectively, both studies observed lower rates of persistent bacteraemia in the fosfomycin groups.

Methods. We will perform a post-hoc analysis of pooled individual patient data from the BACSARM and SAFO trials, which will be referred to as the BACSAFO study. The primary exposure of interest is fosfomycin adjunctive therapy, and the primary outcome will be treatment success at 8 weeks, defined as the patient being alive, without signs of relapse, and showing improvement in clinical signs and symptoms. We will use both Bayesian and frequentist methodologies: the Bayesian analysis will use a hierarchical Bayesian log-binomial model, while the frequentist analysis will apply a hierarchical log-binomial model. In addition, we will investigate whether adjunctive fosfomycin is particularly beneficial in specific patient subgroups (created according to age, methicillin resistance, place of acquisition, and complicated bacteraemia status).

Discussion. The BACSAFO study aims to clarify the role of fosfomycin as an adjunctive therapy for improving outcomes in SAB patients. Although previous trials have not demonstrated significant differences in the primary endpoints, the significant reductions in rates of persistent bacteraemia observed suggest that fosfomycin might offer a clinical benefit in certain cases. By analysing pooled data and attempting to identify subgroups that might benefit most, this study has the potential to refine treatment strategies and inform trial design and planning for future RCTs investigating combination antibiotic therapies for SAB.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the BACSARM and SAFO clinical trials.

Exclusion Criteria:

* For both trials: polymicrobial bacteraemia, severe clinical status with expected survival < 24 hours, severe liver disease with Child-Pugh score class C, diagnosis of prosthetic infective endocarditis, allergy or known resistance to study drugs, pregnancy at the time of inclusion, inclusion in another clinical trial.
* For the BACSARM trial: diagnosis of MRSA pneumonia, prior history of eosinophilic pneumonia, use of additional antibiotic therapy with microbiological activity against MRSA.
* For the SAFO trial: prior history of myasthenia gravis, acute SARS-CoV2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the BACSARM trial, 155 adult patients with MRSA bacteraemia were randomised 1:1 to receive daptomycin in combination with fosfomycin or daptomycin alone. In the SAFO trial, 214 adult patients with MSSA bacteraemia were randomised 1:1 to receive cloxacillin in combination with fosfomycin or cloxacillin alone. As this is a pooled analysis of all SAB, all patients included in the intention-to-treat analysis of the BACSARM and SAFO trials will be included in the present study, regardless of their susceptibility to methicillin.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 8 weeks from the time of randomisation | 8 weeks from the time of randomisation
  A composite outcome available from the information collected in both trials and based on the fulfilment of all the following criteria:
  * Alive at week 8 from the time of randomisation.
  * Absence of relapse within 8 weeks after randomisation, defined as isolation of S. aureus in blood cultures after the index blood cultures were cleared.
  * Improvement of clinical signs and symptoms as assessed by investigators of the BACSARM and SAFO trials at week 8 from the time of randomisation.

SECONDARY OUTCOMES:
Persistent bacteraemia | At days 3 and 7 from the time of randomisation
  Positive blood cultures for S. aureus at days 3 and 7 from the time of randomisation
Mortality at days 14, 30 and 60 from the time of randomisation | Days 14, 30 and 60 from the time of randomisation
  Mortality at days 14, 30 and 60 from the time of randomisation
Adverse events leading to treatment discontinuation | During the time that adjunctive fosfomycin therapy was administered
  Adverse events leading to treatment discontinuation during adjunctive fosfomycin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Carratalà, Medical Doctor, Principal Investigator — Department of Infectious Diseases, Bellvitge University Hospital-IDIBELL, L'Hospitalet de Llobregat, Barcelona, Spain
Locations (6):
- The Royal Melbourne Hospital, at the Peter Doherty Institute for Infection and Immunity, Melbourne, Victoria, Australia
- Institute of Health Policy, Management and Evaluation, University of Toronto, Toronto, Ontario, Canada
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Germans Trias i Pujol Research Institute and Hospital (IGTP), Badalona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
Individual data cannot be shared because of privacy restrictions. Raw anonymised data relating to primary and secondary outcomes and safety can be shared upon request to researchers who provide a methodologically reasonable proposal. The request for data can be sent to the corresponding author (J.C.). A period of 18 months after publication of the main study results should elapse before requests are made, so as to allow authors to publish substudies. Interested researchers must obtain the approval of the Bellvitge University Hospital Ethics Committee.
Supporting Information: Study Protocol, CSR
Time Frame: A period of 18 months after publication of the main study results should elapse before requests are made.
Access Criteria: Researchers who request to BACSAFO principal investigators providing a methodologically reasonable proposal. Interested researchers must obtain the approval of the Bellvitge University Hospital Ethics Committee.

REFERENCES:
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Chow JW, Yu VL. Combination antibiotic therapy versus monotherapy for gram-negative bacteraemia: a commentary. Int J Antimicrob Agents. 1999 Jan;11(1):7-12. doi: 10.1016/s0924-8579(98)00060-0. PMID 10075272
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Grillo S, Pujol M, Miro JM, Lopez-Contreras J, Euba G, Gasch O, Boix-Palop L, Garcia-Pais MJ, Perez-Rodriguez MT, Gomez-Zorrilla S, Oriol I, Lopez-Cortes LE, Pedro-Botet ML, San-Juan R, Aguado JM, Gioia F, Iftimie S, Morata L, Jover-Saenz A, Garcia-Pardo G, Loeches B, Izquierdo-Cardenas A, Goikoetxea AJ, Gomila-Grange A, Dietl B, Berbel D, Videla S, Hereu P, Padulles A, Pallares N, Tebe C, Cuervo G, Carratala J; SAFO study group. Cloxacillin plus fosfomycin versus cloxacillin alone for methicillin-susceptible Staphylococcus aureus bacteremia: a randomized trial. Nat Med. 2023 Oct;29(10):2518-2525. doi: 10.1038/s41591-023-02569-0. Epub 2023 Oct 2. PMID 37783969
- [Background] Pujol M, Miro JM, Shaw E, Aguado JM, San-Juan R, Puig-Asensio M, Pigrau C, Calbo E, Montejo M, Rodriguez-Alvarez R, Garcia-Pais MJ, Pintado V, Escudero-Sanchez R, Lopez-Contreras J, Morata L, Montero M, Andres M, Pasquau J, Arenas MD, Padilla B, Murillas J, Jover-Saenz A, Lopez-Cortes LE, Garcia-Pardo G, Gasch O, Videla S, Hereu P, Tebe C, Pallares N, Sanllorente M, Dominguez MA, Camara J, Ferrer A, Padulles A, Cuervo G, Carratala J; MRSA Bacteremia (BACSARM) Trial Investigators. Daptomycin Plus Fosfomycin Versus Daptomycin Alone for Methicillin-resistant Staphylococcus aureus Bacteremia and Endocarditis: A Randomized Clinical Trial. Clin Infect Dis. 2021 May 4;72(9):1517-1525. doi: 10.1093/cid/ciaa1081. PMID 32725216
- [Background] Garcia-de-la-Maria C, Gasch O, Castaneda X, Garcia-Gonzalez J, Soy D, Canas MA, Ambrosioni J, Almela M, Pericas JM, Tellez A, Falces C, Hernandez-Meneses M, Sandoval E, Quintana E, Vidal B, Tolosana JM, Fuster D, Llopis J, Moreno A, Marco F, Miro JM; Hospital Clinic Endocarditis Study Group. Cloxacillin or fosfomycin plus daptomycin combinations are more active than cloxacillin monotherapy or combined with gentamicin against MSSA in a rabbit model of experimental endocarditis. J Antimicrob Chemother. 2020 Dec 1;75(12):3586-3592. doi: 10.1093/jac/dkaa354. PMID 32853336
- [Background] Kastoris AC, Rafailidis PI, Vouloumanou EK, Gkegkes ID, Falagas ME. Synergy of fosfomycin with other antibiotics for Gram-positive and Gram-negative bacteria. Eur J Clin Pharmacol. 2010 Apr;66(4):359-68. doi: 10.1007/s00228-010-0794-5. Epub 2010 Feb 26. PMID 20186407
- [Background] Garcia-de-la-Maria C, Gasch O, Garcia-Gonzalez J, Soy D, Shaw E, Ambrosioni J, Almela M, Pericas JM, Tellez A, Falces C, Hernandez-Meneses M, Sandoval E, Quintana E, Vidal B, Tolosana JM, Fuster D, Llopis J, Pujol M, Moreno A, Marco F, Miro JM. The Combination of Daptomycin and Fosfomycin Has Synergistic, Potent, and Rapid Bactericidal Activity against Methicillin-Resistant Staphylococcus aureus in a Rabbit Model of Experimental Endocarditis. Antimicrob Agents Chemother. 2018 May 25;62(6):e02633-17. doi: 10.1128/AAC.02633-17. Print 2018 Jun. PMID 29610194
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF; Infectious Diseases Society of America. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children. Clin Infect Dis. 2011 Feb 1;52(3):e18-55. doi: 10.1093/cid/ciq146. Epub 2011 Jan 4. PMID 21208910
- [Background] Paul M, Zemer-Wassercug N, Talker O, Lishtzinsky Y, Lev B, Samra Z, Leibovici L, Bishara J. Are all beta-lactams similarly effective in the treatment of methicillin-sensitive Staphylococcus aureus bacteraemia? Clin Microbiol Infect. 2011 Oct;17(10):1581-6. doi: 10.1111/j.1469-0691.2010.03425.x. Epub 2010 Dec 14. PMID 21073629
- [Background] GBD 2021 Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance 1990-2021: a systematic analysis with forecasts to 2050. Lancet. 2024 Sep 28;404(10459):1199-1226. doi: 10.1016/S0140-6736(24)01867-1. Epub 2024 Sep 16. PMID 39299261
- [Background] Gasch O, Camoez M, Dominguez MA, Padilla B, Pintado V, Almirante B, Molina J, Lopez-Medrano F, Ruiz E, Martinez JA, Bereciartua E, Rodriguez-Lopez F, Fernandez-Mazarrasa C, Goenaga MA, Benito N, Rodriguez-Bano J, Espejo E, Pujol M; REIPI/GEIH Study Groups. Predictive factors for mortality in patients with methicillin-resistant Staphylococcus aureus bloodstream infection: impact on outcome of host, microorganism and therapy. Clin Microbiol Infect. 2013 Nov;19(11):1049-57. doi: 10.1111/1469-0691.12108. Epub 2013 Jan 17. PMID 23331461
- [Background] Kuehl R, Morata L, Boeing C, Subirana I, Seifert H, Rieg S, Kern WV, Kim HB, Kim ES, Liao CH, Tilley R, Lopez-Cortes LE, Llewelyn MJ, Fowler VG, Thwaites G, Cisneros JM, Scarborough M, Nsutebu E, Gurgui Ferrer M, Perez JL, Barlow G, Hopkins S, Ternavasio-de la Vega HG, Torok ME, Wilson P, Kaasch AJ, Soriano A; International Staphylococcus aureus collaboration study group and the ESCMID Study Group for Bloodstream Infections, Endocarditis and Sepsis. Defining persistent Staphylococcus aureus bacteraemia: secondary analysis of a prospective cohort study. Lancet Infect Dis. 2020 Dec;20(12):1409-1417. doi: 10.1016/S1473-3099(20)30447-3. Epub 2020 Aug 4. PMID 32763194
- [Background] Minejima E, Mai N, Bui N, Mert M, Mack WJ, She RC, Nieberg P, Spellberg B, Wong-Beringer A. Defining the Breakpoint Duration of Staphylococcus aureus Bacteremia Predictive of Poor Outcomes. Clin Infect Dis. 2020 Feb 3;70(4):566-573. doi: 10.1093/cid/ciz257. PMID 30949675
- [Background] Inagaki K, Lucar J, Blackshear C, Hobbs CV. Methicillin-susceptible and Methicillin-resistant Staphylococcus aureus Bacteremia: Nationwide Estimates of 30-Day Readmission, In-hospital Mortality, Length of Stay, and Cost in the United States. Clin Infect Dis. 2019 Nov 27;69(12):2112-2118. doi: 10.1093/cid/ciz123. PMID 30753447
- [Background] Stewardson AJ, Allignol A, Beyersmann J, Graves N, Schumacher M, Meyer R, Tacconelli E, De Angelis G, Farina C, Pezzoli F, Bertrand X, Gbaguidi-Haore H, Edgeworth J, Tosas O, Martinez JA, Ayala-Blanco MP, Pan A, Zoncada A, Marwick CA, Nathwani D, Seifert H, Hos N, Hagel S, Pletz M, Harbarth S; TIMBER Study Group. The health and economic burden of bloodstream infections caused by antimicrobial-susceptible and non-susceptible Enterobacteriaceae and Staphylococcus aureus in European hospitals, 2010 and 2011: a multicentre retrospective cohort study. Euro Surveill. 2016 Aug 18;21(33):30319. doi: 10.2807/1560-7917.ES.2016.21.33.30319. PMID 27562950
- [Background] Kaasch AJ, Barlow G, Edgeworth JD, Fowler VG Jr, Hellmich M, Hopkins S, Kern WV, Llewelyn MJ, Rieg S, Rodriguez-Bano J, Scarborough M, Seifert H, Soriano A, Tilley R, Torok ME, Weiss V, Wilson AP, Thwaites GE; ISAC, INSTINCT, SABG, UKCIRG, and Colleagues. Staphylococcus aureus bloodstream infection: a pooled analysis of five prospective, observational studies. J Infect. 2014 Mar;68(3):242-51. doi: 10.1016/j.jinf.2013.10.015. Epub 2013 Nov 16. PMID 24247070
- [Background] IHME Pathogen Core Group. Global burden associated with 85 pathogens in 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Infect Dis. 2024 Aug;24(8):868-895. doi: 10.1016/S1473-3099(24)00158-0. Epub 2024 Apr 16. PMID 38640940
- [Background] Diekema DJ, Hsueh PR, Mendes RE, Pfaller MA, Rolston KV, Sader HS, Jones RN. The Microbiology of Bloodstream Infection: 20-Year Trends from the SENTRY Antimicrobial Surveillance Program. Antimicrob Agents Chemother. 2019 Jun 24;63(7):e00355-19. doi: 10.1128/AAC.00355-19. Print 2019 Jul. PMID 31010862
- [Background] Martinez Perez-Crespo PM, Lopez-Cortes LE, Retamar-Gentil P, Garcia JFL, Vinuesa Garcia D, Leon E, Calvo JMS, Galan-Sanchez F, Natera Kindelan C, Del Arco Jimenez A, Sanchez-Porto A, Herrero Rodriguez C, Becerril Carral B, Molina IMR, Iglesias JMR, Perez Camacho I, Guzman Garcia M, Lopez-Hernandez I, Rodriguez-Bano J; PROBAC REIPI/GEIH-SEIMC/SAEI Group. Epidemiologic changes in bloodstream infections in Andalucia (Spain) during the last decade. Clin Microbiol Infect. 2021 Feb;27(2):283.e9-283.e16. doi: 10.1016/j.cmi.2020.05.015. Epub 2020 May 26. PMID 32470569
- [Derived] Escrihuela-Vidal F, Ong SWX, Oriol I, Grillo S, Pujol M, Pallares N, Tebe C, Liu K, Miro JM, Tong SYC, Carratala J. Adjunctive Fosfomycin for the Treatment of Staphylococcus aureus Bacteremia: A Pooled Post-hoc Analysis of Individual Participant Data from Two Randomized Trials. Clin Infect Dis. 2025 Jul 16:ciaf387. doi: 10.1093/cid/ciaf387. Online ahead of print. PMID 40670317